CLINICAL TRIAL: NCT03092362
Title: Beat-to-beat Variability in Persistent Atrial Fibrillation
Acronym: BVAR-Afib
Status: Completed | Type: Observational
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Sponsor
Other Study IDs: HDZNRW-KA-009-HO
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-07

CONDITIONS: Persistent Atrial Fibrillation
Keywords: persistent atrial fibrillation; Heart rate variability; quality of life
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Heart rate variability (HRV) in patients with atrial fibrillation (AF) is hardly studied. Though a reduced HRV in patients with heart failure and reduced ejection fraction (HFrEF) has been associated with poor prognosis. Data on HRV in AF-patients without a reduced ejection fraction is lacking. We hypothesize that those patients with persistent atrial fibrillation and larger beat-to-beat variability would be more symptomatic than does those with smaller HRV. To asses this theory we intend to perform a prospective observational trial. Symptoms of Atrial fibrillation will be assessed using Quality of Life questionnaires and 6 minutes walking test. Heart rate variability will be assessed using 24 hour Holter ECG monitoring.

The correlation between symptoms and heart rate variability will be then assessed.

ELIGIBILITY:
Inclusion Criteria:

* Persistent atrial fibrillation
* No previous ablation for atrial fibrillation
* At least 18 years old
* Signed written patient's informed consent

Exclusion Criteria:

* Paroxysmal atrial fibrillation
* Previous ablation therapy for atrial fibrillation
* Reduced left ventricular ejection fraction (LVEF<35%)
* Permanent ventricular pacing (including cardiac resynchronization therapy CRT)
* Acute coronary syndrome (ACS) during past 6 weeks.
* Stroke or TIA within past 6 weeks.
* Cardiac surgical operation/ intervention within past 3 months.
* Acute decompensated heart failure
* Treatment with IV Inotropic medications (e.g. Dobutamine, Levosimendan)
* Mitral valve replacement or rheumatic mitral valve stenosis
* Neurological or psychological disease that may impair patient's judgement or compliance
* Pregnancy or Breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with persistent atrial fibrillation (defined as lasting more than seven days or requiring termination by cardioversion either with drugs or by direct current cardioversion) who are admitted at our clinic.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-11; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation symptoms | 7 days
  Whether atrial fibrillation symptoms assessed by Quality-of-Life questionnaires correlates with heart rate variability

SECONDARY OUTCOMES:
Atrial fibrillation symptoms | 7 days
  Whether atrial fibrillation symptoms assessed by Quality-of-Life questionnaires correlates with heart rate reserve. Heart rate reserve is defined as the difference between maximal heart rate (220- age in years) and mean heart rate during atrial fibrillation (assessed by 24 hour Holter ECG monitoring).
Improvement in 6MWD (6 minutes walk distance) | 7 days
  Whether 6MWD improvement after treatment of atrial fibrillation correlates with heart rate variability.

CONTACTS AND LOCATIONS:
Overall Officials: Hazem Omran, MD, Principal Investigator — HDZ NRW
Locations (1):
- Heart and Diabetes Center NRW, Bad Oeynhausen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cygankiewicz I, Corino V, Vazquez R, Bayes-Genis A, Mainardi L, Zareba W, de Luna AB, Platonov PG; MUSIC Trial Investigators. Reduced Irregularity of Ventricular Response During Atrial Fibrillation and Long-term Outcome in Patients With Heart Failure. Am J Cardiol. 2015 Oct 1;116(7):1071-5. doi: 10.1016/j.amjcard.2015.06.043. Epub 2015 Jul 16. PMID 26298305